CLINICAL TRIAL: NCT01968785
Title: RENAL ARTERY IRRADIATION FOR SYMPATHETIC RENAL DENERVATION IN PATIENTS WITH RESISTANT HYPERTENSION
Brief Title: Renal Denervation in Patients With Uncontrolled Blood Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Renal Denervation
Record Dates: First submitted 2013-10-16; First posted 2013-10-24 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiation dose 25 Gy (Active Comparator): • 25 Gy: Subjects will be treated with beta radiation dosage of 25 Gy during renal denervation procedure. Subjects are to maintain baseline anti-hypertensive medications and will undergo follow-up for 24 months.
  Interventions: Radiation: Radiation Dose 25 Gy
- Radiation dose 50 Gy (Active Comparator): • 50 Gy: Subjects will be treated with beta radiation dosage of 50 Gy during renal denervation procedure. Subjects are to maintain baseline anti-hypertensive medications and will undergo follow-up for 24 months.
  Interventions: Radiation: Radiation Dose 50 Gy

INTERVENTIONS:
Radiation: Radiation Dose 25 Gy — Renal Denervation is performed using the Beta-Cath 3.5F to a deliver radiation dose 25 Gy to the renal artery.
  Arms: Radiation dose 25 Gy
Radiation: Radiation Dose 50 Gy — Renal Denervation is performed using the Beta-Cath 3.5F to a deliver radiation dose 50 Gy to the renal artery.
  Arms: Radiation dose 50 Gy

SUMMARY:
The kidneys are an important regulator of blood pressure. Previous research has shown that disrupting the nerves (denervate) of the kidney may successfully decrease blood pressure. In the past, one technique that was used to treat severe high blood pressure was a surgical procedure to cut these nerves. However, this surgery is no longer commonly performed.

Another approach to disrupting these nerves is to use the Beta-Cath 3.5F system to deliver a small amount of radiation to the treatment zone. The Beta-Cath 3.5F System (Novoste) is currently approved in the United States to deliver ion dose therapy to re-narrowings that form in the coronary arteries in the heart. This trial is assessing the safety of treating patients with the Beta-Cath 3.5F System (Novoste) to denervate the nerves around the kidney to help control blood pressure in patients with uncontrolled hypertension.

1. Renal artery brachytherapy with beta-emitting source is safe.
2. Renal artery brachytherapy with beta-emitting source can reduce systolic/diastolic blood pressure via renal denervation mechanism within 6 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* 4.2.1 GENERAL INCLUSION CRITERIA

Subjects must meet all of the following inclusion criteria prior to enrollment into the trial:

1. Individual is ≥ 18 and ≤ 85 years of age.
2. Individual has a systolic blood pressure (SBP) ≥ 160 mmHg (≥ 150 mmHg for type 2 diabetics) based on an average of 3 office blood pressure readings.
3. Individual is adhering to a stable (maximally tolerated dose) drug regimen including 3 or more anti-hypertensive medications for at least 1 month (including one diuretic) that is expected to be maintained for at least 6 months.
4. Individual is competent and willing to provide informed consent to participate in the trial.

4.2.2 ANGIOGRAPHIC INCLUSION CRITERIA

1. Individual has main renal arteries measuring <2.75 mm in diameter.

Exclusion Criteria:

1. Inability to sign written informed consent.
2. Individual has renal artery anatomy that is ineligible for treatment including:

   1. Main renal arteries with <20 mm treatable length
   2. Renal artery stenosis of ≥20% by angiography.
   3. A history of prior renal artery intervention including balloon angioplasty or stenting.
   4. Multiple main renal arteries in either kidney.
3. Individual has an eGFR of < 45mL/min/1.73m2, using the MDRD formula calculation.
4. Individual has had >1 hospital admission for a hypertensive crisis within the past year.
5. Individual has an Ambulatory Blood Pressure Monitoring 24 hour average SBP<135mmHg.
6. Individual has has > 1 episode(s) of orthostatic hypotension (reduction of SBP of >20 mmHg or diastolic blood pressure (DBP) of >10 mmHg within 3 minutes of standing) coupled with symptoms within the past year or during the screening process.
7. Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
8. Individual has primary pulmonary hypertension.
9. Individual has scheduled or planned surgery or cardiovascular intervention in the next 3 months.
10. Individual has a condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement using the protocol-specified automatic blood pressure monitor (e.g., arm diameter too large for the cuff, arrhythmia that interferes with automatic monitor's pulse sensing and prohibits an accurate measurement).
11. Individual is pregnant, nursing or planning to be pregnant.
12. Individual has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
13. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia, or arrhythmias such as atrial fibrillation).
14. Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
15. Individual is currently enrolled in another investigational drug or device trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: no patients were enrolled in arm two
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety-renal Artery Brachytherapy With Beta-emitting Source is Any Need for Renal Artery Intervention to Treat Renal Artery Injury Induced by the Catheter of Radiation Within 6 Months
Description: The primary safety endpoint for renal artery brachytherapy with beta-emitting source is any need for renal artery intervention to treat renal artery injury induced by the catheter of radiation within 6 months
Time Frame: up to 6 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Efficacy- Renal Artery Brachytherapy With Beta-emitting Source is Decrease in Systolic and Diastolic Blood Pressure of ≥10 mmHg at Six Months Following the Procedure.
Description: The primary efficacy endpoint for renal artery brachytherapy with beta-emitting source is decrease in systolic and diastolic blood pressure of ≥10 mmHg at six months following the procedure.
Time Frame: up to 6 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Angiographic
Description: The angiographic endpoint is defined as late loss at 6 months by offline quantitative coronary angiography (QCA)
Time Frame: up to 6 months post procedure
Population: not enough patients were enrolled to analize data
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Effects on Blood Pressure
Description: Short term effects of renal artery brachytherapy on blood pressure
Time Frame: up to 6 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Safety-renal Artery Dissection or Perforation Requiring Intervention, and Serious Groin Complications Specifically.
Description: Acute procedural safety; renal artery dissection or perforation requiring intervention, and serious groin complications specifically.
Time Frame: up to 24 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: eGFR or New Stenosis
Description: Estimated glomerular filtration rate (eGFR) drop >25% or new renal artery stenosis > 60% confirmed by angiogram at six months following renal artery brachytherapy procedure.
Time Frame: up to 6 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Medication Changes
Description: Any changes made in the patients' blood pressure medication regimen throughout the 24 month duration. Specifically,
  1. Additions, changes and cessation of medications
  2. Dosage changes throughout the follow up duration
Time Frame: up to 24 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Serious Adverse Events
Description: Rate of any serious adverse events or device-related adverse events
Time Frame: up to 24 months post procedure
Population: Not enough patients were enrolled to be analyzed
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Radiation Dose 50 Gy: No patients were enrolled in this arm of the study
Arm/Group | Radiation Dose 25 Gy | Radiation Dose 50 Gy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Dose 25 Gy (N=2) | Radiation Dose 50 Gy (N=0)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes